CLINICAL TRIAL: NCT04045561
Title: Elaboration of a Standardized Referential Guide of the Information to Optimize the Adherence to be Given During an Initial Pharmaceutical Consultation (CP) to the Patient Suffering From Multiple Myeloma in Primocure Chemotherapy Per os
Brief Title: Development of a Standardized Reference Guide for Tuning Adherence to Dispense During a Initial Pharmaceutical Consulting (CP ) to the Patient With Multiple Myeloma Oral Chemotherapy Primocure
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2015/MF-01
Record Dates: First submitted 2019-07-23; First posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The hypothesis is that the implementation of an initial Pharmaceutical Consultation (PC) program based on the provision of standardized information to patients treated for multiple myeloma as a first course of chemotherapy, could optimize their compliance with the delivered per os treatment.

The aim of this study is therefore to develop a standardised reference guide of information to be provided during prostate cancer in order to optimise the compliance of patients treated for multiple myeloma as a first course of chemotherapy per os.

ELIGIBILITY:
Inclusion criteria

* The patient must be a member or beneficiary of a health insurance plan
* The patient is at least 18 years old
* The patient is treated for multiple myeloma, is naive to any treatment and begins a chemotherapy protocol with oral therapy and whose course of care includes a stay in the Day Hospital or retrocessions.

Criteria for non-inclusion

* The subject is participating in another study
* The subject is in an exclusion period determined by a previous study
* The subject is under the protection of justice, guardianship or curatorship
* It is impossible to give informed information about
* The patient is pregnant, parturient, or breastfeeding
* The patient receives a follow-up by a home nurse for the administration of oral medication
* The patient is treated only with oral chemotherapy in the city
* The patient has early dementia.

Translated with www.DeepL.com/Translator

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient is treated for multiple myeloma, is naive to any treatment and begins a chemotherapy protocol with oral therapy and whose course of care includes a stay in the Day Hospital or retrocessions.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
evaluating the understanding | Day 1
  Questionnaire. quantitative variables: measurement of the mean and standard deviation or by their median and quartiles according to their distribution.
evaluating understanding | Day 1
  Questionnaire. qualitative variables: measurement of their number and
evaluating the quality of information | Day 1
  Questionnaire. quantitative variables: measurement of the mean and standard deviation or by their median and quartiles according to their distribution.
evaluating quality of information | Day 1
  Questionnaire. qualitative variables: measurement of their number and percentage.

SECONDARY OUTCOMES:
The time required for the pharmaceutical consultation | Day 1
  minutes
satisfaction des patients | Day 1
  by an Analogue Visual Scale (0-10-very satisfied)